CLINICAL TRIAL: NCT05271227
Title: Assessment Of Volume Responsiveness By Ultrasound Parameters Of Carotid Blood Flow In Patients With Cardiogenic Shock
Brief Title: Volume Responsiveness By Ultrasound Of Carotid Blood Flow In Patients With Cardiogenic Shock
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nehal Yousri, Resident physician at AMUH, Principal investigator, MD student, Alexandria University
Other Study IDs: VR by CBF in CS patients
Record Dates: First submitted 2022-01-23; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Cardiogenic Shock; Volume Responsiveness; Ultrasound
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiogenic Shock Patients: Cardiac output and Carotid Blood flow is measured before & after PLR test, then percent change is calculated were increase in cardiac output with 10 % or more is considered volume responder.
  Measurements can be repeated as needed, and fluid resuscitation continues until no further response to passive leg raising is noted.
  Interventions: Other: Transthoracic echocardiography and Carotid artery doppler (PHILIPS HD11 XE ultrasound device) before and after PLR test.

INTERVENTIONS:
Other: Transthoracic echocardiography and Carotid artery doppler (PHILIPS HD11 XE ultrasound device) before and after PLR test. — VTI-LVOT was measured by echo by placing the pulsed wave Doppler sample gate in the LVOT diameter in apical-5-chamber window. VTI-LVOT was obtained by manually tracing the Doppler velocity spectrum. LVOT velocity time integral was recorded before and after PLR test within 2 minutes. Carotid blood flow was measured by using two-dimensional image, the optimal image of the long-axis view was obtained at the common carotid artery. The sample volume was placed on the center of the lumen, 2 cm proximal to the bulb, and a pulsed wave Doppler examination,The angle correction cursor was placed parallel to the direction of blood flow. A PLR will be performed in 2 sequential steps, first step patient is seated in the semi recumbent position (45°) then using an automatic bed elevation technique, the lower limbs will be then raised to a 45° angle while the patient's trunk will be lowered in supine position. Thus, the angle between the trunk and the lower limbs will remain unchanged (135°).

SUMMARY:
Resuscitation of critically ill patients has changed since the advent of goal directed therapy. Today, practitioners providing fluid resuscitation are attentive of the danger associated with volume depletion while being aware of the morbidity of volume overload. Fluid resuscitation must be rapid, precise, and individually tailored to each patient based on reliable data obtained by various means inside ICU setting.

There is no non-invasive method that can reliably and accurately identify fluid responsiveness. As such, in patients with undifferentiated shock, treatment often involves empiric fluid administration, in the hopes that volume expansion will increase preload, which will then serve to increase cardiac output (CO). However, for patients on the flat portion of the Starling curve, aggressive fluid administration results in no appreciable increase in CO and may be detrimental to hemodynamically unstable patients.

DETAILED DESCRIPTION:
Study location and population: Alexandria Main University Hospitals ICU, Alexandria Egypt. Approval of the Medical Ethics Committee of Alexandria Faculty of Medicine was obtained before the start of the study. Sample size was estimated using PASS version 20 program. The minimal hypothesized total sample size of 40 cardiogenic shock patients of both sexes is needed to determine the sensitivity and specificity of cardiac output measurement using either bedside ultrasound on carotid artery and TTE (Standard) while assessing volume responsiveness with 95 % confidence level and 80 % power using z-test.

Study procedures: All enrolled patients were subjected on admission to thorough history taking including age, sex, date of ICU admission and preexisting underlying disease (Diabetes Mellitus, hypertension), presence of sepsis, smoking, analgesic abuse. Full clinical examination. Severity of illness was assessed by Acute Physiological And Chronic Health Evaluation-ΙΙ (APACHE ΙΙ). ICU length of stay (LOS) and final outcome were recorded.

Noninvasive measurement of Systolic arterial pressure, diastolic arterial pressure (DAP), mean arterial pressure (MAP), heart rate (HR), respiratory rate (RR), and temperature were recorded upon admission and after PLR.

Fluid challenge: A PLR was performed, Transferring a patient to the passive leg raising (PLR) position (in which the lower limbs are elevated at 45_ while the trunk is lying supine) transfers venous blood from the legs to the intrathoracic compartment and increases cardiac preload around 300-500 mL.

Carotid ultrasonography and Echocardiogram: Stroke volume is the amount of blood ejected from the ventricle with each cardiac cycle. It can be readily calculated by subtracting the end-systolic volume from the end-diastolic volume. Multiplying the stroke volume by the heart rate yields the cardiac output, typically reported in liters per minute.

Stroke volume can be estimated by using a combination of 2D and Doppler imaging. HR was recorded before and after PLR test then CO is calculated by equation of:

CO = π × (LVOTd)2/4 × VTI LVOT × HR Percent change is [(cardiac output after passive leg raising - cardiac output before passive leg raising)/cardiac output after passive leg raising] × 100%. A greater than 10% increase in cardiac output would predict volume responsiveness and constitute an indication for a 500-mL fluid bolus. Measurements were repeated as needed, and fluid resuscitation continued until no further response to passive leg raising was noted.

Changes (%) =100 X (post-FC value - baseline value)/ baseline value

Patients were divided into 2 groups:

Responder is defined by an increase of 10% or more. Non responder is less than 10%. The Common Carotid artery is a large superficial accessible artery so carotid doppler flow imaging would be simple, non-invasive method to assess volume responsiveness. Use of Velocity Time Integral of flow through the Common Carotid artery (Carotid VTI) and Passive Leg Raising (PLR) described as a marker of volume responsiveness in hemodynamically unstable patients.

Carotid flow is measured during the passive leg raising maneuver by using a linear array transducer positioned in the long axis over the CCA, after procuring a longitudinal view of the common carotid artery, pulsed Doppler analysis at 2 cm from the bifurcation was performed. The CCA diameter is measured from opposing points of the vessel's intimal wall, with the velocity time integral determined automatically using spectral Doppler envelopes and the sample obtained from the center of the artery. Common carotid artery blood flow per minute is calculated by the equation CBF= π × (CCA diameter)2/4 × CCA velocity time integral × heart rate This parameter is measured both before and after the passive leg raising to determine the percent change in CCA blood flow. An increase in CCA flow with passive leg raising only occurs in patients with shock, and an increase of greater than 20% is highly predictive of volume responsiveness.

HR is recorded before and after PLR then CBF was calculated by the following equation:

CBF = π × (CCA diameter)2/4 × VTI CCA × HR

Patients was divided into 2 groups:

Responder is defined by an increase of 20% or more. Non responder is less than 20%. After fluid challenge we remeasured Systolic arterial pressure, diastolic arterial pressure (DAP), mean arterial pressure (MAP), heart rate (HR) to assess clinical response to the fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Y.
* Cardiogenic shock.

Exclusion Criteria:

* Age < 18 Y.
* Pregnant females.
* All types of shock state other than cardiogenic.
* Peripheral arterial disease.
* Non consenting patients.
* Unable to tolerate passive leg raise (PLR).
* Common carotid artery stenosis greater than 50 % (systolic peak velocity >182 cm/s and/or diastolic velocity >30 cm/s by Doppler ultrasound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 cardiogenic shock patients of both gender admitted to intensive critical care units.
  Approval of the Medical Ethics Committee of Alexandria Faculty of Medicine. An informed consent was taken from the patients' next of kin before their enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Percent Change in Carotid Blood Flow after PLR test. | Change in carotid blood flow within 2 minutes after PLR.
  The common carotid artery will be scanned in transverse and longitudinal planes. Spectral Doppler tracings will be then obtained by placing a 0.5 mm sample gate through the center of vessel, within 2-3 cm proximal to the carotid bulb in the longitudinal plane, in accordance to standard guidelines. The angle correction cursor will be placed parallel to the direction of blood flow. A PLR will be performed in 2 sequential steps, first step patient is seated in the semi recumbent position (45°) then using an automatic bed elevation technique, the lower limbs will be then raised to a 45° angle while the patient's trunk will be lowered in supine position. Thus, the angle between the trunk and the lower limbs will remain unchanged (135°). Percent change is [(cardiac output after passive leg raising - carotid blood flow before passive leg raising)/carotid blood flow after passive leg raising] × 100%. A greater than 20% increase in carotid blood flow would predict volume responsiveness.
Percent Change in Cardiac Output after PLR test. | Change in cardiac output within 2 minutes after PLR.
  Cardiac output is measured using pulsed Doppler imaging where phase-array transducer positioned just proximal to the aortic valve. The velocity time integral is measured by tracing the modal velocity then stroke volume is calculated.CO is SV multiplied by HR. A PLR will be performed in 2 sequential steps, first step patient is seated in the semi recumbent position (45°) then using an automatic bed elevation technique, the lower limbs will be then raised to a 45° angle while the patient's trunk will be lowered in supine position. Thus, the angle between the trunk and the lower limbs will remain unchanged (135°). Percent change is [(cardiac output after passive leg raising - cardiac output before passive leg raising)/cardiac output after passive leg raising] × 100%. A greater than 10% increase in cardiac output would predict volume responsiveness.
Blood Pressure before and after PLR test. | Change in blood pressure 1 minute after PLR.
  Measure Blood Pressure and record reading in mmHg before and after PLR test.
Heart rate before and after PLR test. | Change in heart rate 1 minute after PLR.
  Record Heart Rate readings on monitor in BPM (beat per minute) before and after PLR test.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M ElMenshawy, Lecturer, Study Director — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Sadaka F, Juarez M, Naydenov S, O'Brien J. Fluid resuscitation in septic shock: the effect of increasing fluid balance on mortality. J Intensive Care Med. 2014 Jul-Aug;29(4):213-7. doi: 10.1177/0885066613478899. Epub 2013 Feb 27. PMID 23753235
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Evans D, Ferraioli G, Snellings J, Levitov A. Volume responsiveness in critically ill patients: use of sonography to guide management. J Ultrasound Med. 2014 Jan;33(1):3-7. doi: 10.7863/ultra.33.1.3. No abstract available. PMID 24371093
- [Background] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Background] Ma IWY, Caplin JD, Azad A, Wilson C, Fifer MA, Bagchi A, Liteplo AS, Noble VE. Correlation of carotid blood flow and corrected carotid flow time with invasive cardiac output measurements. Crit Ultrasound J. 2017 Dec;9(1):10. doi: 10.1186/s13089-017-0065-0. Epub 2017 Apr 20. PMID 28429291
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963